CLINICAL TRIAL: NCT04708028
Title: Animal Assisted Therapy's Effects on Dental Patients
Brief Title: Animal Assisted Therapy in Dentistry
Acronym: AAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-1911
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No exposure to the therapy dog.
- Dog Therapy (Experimental): Introduced to a therapy dog and allowed to pet the dog for up to 2 minutes (timed) prior to the dental procedure.
  Interventions: Other: Dog Therapy

INTERVENTIONS:
Other: Dog Therapy — The intervention is a therapy dog interaction (e.g. petting) for up to 2 minutes before their appointment and first interaction with the doctor. The subject can pet the dog for as long as they like up until the 2 minute mark.
  Arms: Dog Therapy

SUMMARY:
A cross-sectional prospective study measuring physiologic biometrics and perceptions of stress during a dental procedure with or without a therapy dog present.

DETAILED DESCRIPTION:
Patients will be consented, enrolled, and assigned to a control group (no dog) or to an experimental group (dog). The patient assigned to the experimental group will be exposed to the therapy animal prior to the dental appointment. Pre-dental procedure and post-dental procedure surveys will be given to all the subjects asking the same questions. Biometric data will be collected by measuring heart rates of the patient/subject during the dental appointment with a Shimmer or Polar device.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

* 7-17 years of age
* Patient undergoing 1 quadrant restorative dental procedure requiring a handpiece (e.g. multiple fillings, sealants and/or stainless-steel crowns) and/or extraction(s)
* History of moderate dental anxiety with a Frankl score of 2-3 based on Epic chart review

Exclusion Criteria Subjects presenting with any of the following will not be included in the study:

* Patients with developmental delay/special needs, Autism Spectrum Disorders (ASDs), craniofacial defects, chronic pain conditions, and/or dental syndromes
* No history of dental anxiety
* Moderate to severe allergy to dogs
* Previous traumatic experience with a dog and/or self-reported fear of dogs
* Patients who are not receiving dental care requiring a handpiece (for ex, prophylaxis only)
* Patients with severe, documented xerostomia
* Patients receiving sedation (pharmacological and conscious sedation) or general anesthesia
* Patients who will have physical restraints placed during the dental procedure
* Patient scheduled to have sedation or general anesthesia
* Severe acute or chronic medical or psychiatric condition(s) that would interfere with the interpretation of results, and in the judgement of the Investigator, would make the subject inappropriate for entry into the trial
* Patient with developmental/cognitive disability that cannot self-assent, comprehend and follow the requirements of the study based on research site personnel's assessment.
* Inability or unwillingness of individual and legal guardian/representative to give written informed assent (from child) and consent (from adult).

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2024-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Jacox, DMD, PhD, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- General & Oral Health Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning following publication up to 1 year provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 1 month following publication up to 1 year
Access Criteria: Deidentified individual data that supports the results will be shared beginning following publication up to 1 year provided the investigator who proposes to use the data has approval from an IRB, IEC, or REB as applicable, and an executed data use/sharing agreement with University of North Carolina (UNC).

REFERENCES:
- [Derived] Massouda J, Ghaltakhchyan N, Judd J, Bocklage C, Selden R, TumSuden O, Nanney E, Lee J, Ginnis J, Strauman T, Sawicki C, Hodges EA, Graves C, Divaris K, Jacox L. Evaluating effects of animal-assisted therapy on pediatric dental care patients: A pilot clinical trial. J Am Dent Assoc. 2025 Jun;156(6):447-457.e14. doi: 10.1016/j.adaj.2025.03.006. PMID 40467121

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Dog Therapy
Started | 22 | 18
Completed | 21 | 18
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Dog Therapy | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 18 | 39
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (2.0) | 9.2 (2.1) | 9.6 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 4 | 2 | 6
  More than one race | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Salivary Amylase Levels Throughout Dental Visit
Description: To measure stress levels salivette swab will be placed in child's cheek to absorb saliva.
Time Frame: Up to end of dental visit; a total average between 60 to 90 minutes
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Control | Dog Therapy
Number analyzed (Participants) | 21 | 18
U/mL
  Baseline | 150.82 (135.01) | 166.70 (114.32)
  8 minutes Post intervention (Dog exposure or no dog exposure) | 127.77 (92.46) | 145.39 (99.02)
  8 minutes after starting dental procedure | 97.78 (59.65) | 175.11 (144.37)
  8 minutes after completion of dental procedure | 175.10 (232.24) | 210.05 (188.93)
Statistical Analysis 1: Comparison: Control vs Dog Therapy; Baseline; Test type: Superiority; p = 0.379, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Dog Therapy; 8 minutes Post intervention (Dog exposure or no dog exposure); Test type: Superiority; p = 0.646, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Dog Therapy; 8 minutes after starting dental procedure; Test type: Superiority; p = 0.219, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Dog Therapy; 8 minutes after completion of dental procedure; Test type: Superiority; p = 0.223, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Mean Salivary Cortisol Levels Throughout Dental Visit
Description: To measure stress levels salivette swab will be placed in child's cheek to absorb saliva.
Time Frame: Up to end of dental visit; a total average between 60 to 90 minutes
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | Control | Dog Therapy
Number analyzed (Participants) | 21 | 18
µg/dL
  Baseline | 0.185 (0.255) | 0.155 (0.090)
  8 minutes Post intervention (Dog exposure or no dog exposure) | 0.153 (0.219) | 0.154 (0.112)
  8 minutes after starting dental procedure | 0.223 (0.273) | 0.133 (0.129)
  8 minutes after completion of dental procedure | 0.186 (0.157) | 0.193 (0.127)
Statistical Analysis 1: Comparison: Control vs Dog Therapy; Baseline; Test type: Superiority; p = 0.410, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Control vs Dog Therapy; 8 minutes Post intervention (Dog exposure or no dog exposure); Test type: Superiority; p = 0.127, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Control vs Dog Therapy; 8 minutes after starting dental procedure; Test type: Superiority; p = 0.268, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Control vs Dog Therapy; 8 minutes after completion of dental procedure; Test type: Superiority; p = 0.353, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent for this single visit study through post visit survey collection, a total average between 60 to 90 minutes.
Arm/Group | Control | Dog Therapy
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT04708028/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT04708028/ICF_001.pdf